CLINICAL TRIAL: NCT03292458
Title: Central Mechanisms and Treatment Response of Sodium Oxybate in Spasmodic Dysphonia and Voice Tremor
Brief Title: Sodium Oxybate in Spasmodic Dysphonia and Voice Tremor
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Kristina Simonyan (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor-Investigator, Kristina Simonyan, Professor of Otolaryngology - Head & Neck Surgery, Director of Laryngology Research, Massachusetts Eye and Ear Infirmary
Organization: Massachusetts Eye and Ear Infirmary (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 2019P001680; R01DC012545 (NIH)
Record Dates: First submitted 2017-09-20; First posted 2017-09-25 (Actual); Results first posted 2025-04-04 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Spasmodic Dysphonia; Voice Tremor
Keywords: spasmodic dysphonia; laryngeal dystonia; functional MRI; Xyrem
MeSH Terms: conditions — Dysphonia | interventions — Sodium Oxybate; Ethanol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Clinical response to sodium oxybate (Experimental): In contrast to placebo but similar to alcohol, sodium oxybate is expected to be most effective in reducing voice symptoms in alcohol-responsive SD and VT.
  Interventions: Drug: Sodium Oxybate
- Central markers of clinical response (Experimental): The clinical outcome is expected to be determined by selective modulation of functional abnormalities in the brain regions controlling speech sensorimotor processing and integration in association with underlying gene variants.
  Interventions: Drug: Sodium Oxybate

INTERVENTIONS:
Drug: Sodium Oxybate — Alcohol challenge test and oral administration of a single dose of sodium oxybate and the matching placebo.
  Other Names: Placebo; Alcohol

SUMMARY:
Using a comprehensive approach of clinico-behavioral testing, neuroimaging and pharmacogenetics, the researchers will examine the clinical effects of sodium oxybate and the matched placebo on voice symptoms in spasmodic dysphonia and voice tremor.

DETAILED DESCRIPTION:
Spasmodic dysphonia (SD), or laryngeal dystonia, is a chronic debilitating condition that selectively affects speech production due to involuntary spasms in the laryngeal muscles. SD often extends beyond the impairment of vocal communication causing significant occupational disability and life-long social isolation. SD becomes even more incapacitating when it is associated with dystonic voice tremor (VT), which is present in about 1/3 of SD patients and is characterized by the inability to sustain a vowel for more than a few seconds. Current treatment of these disorders is limited to the temporary management of voice symptoms with repeated injections of botulinum toxin into the laryngeal muscles. These injections, however, are not fully effective in all SD patients and even less so in combined SD and VT cases. There is, therefore, a critical need to identify alternative therapeutic options that specifically target the pathophysiology of these disorders. On the other hand, the design and the use of such novel therapeutic approaches will be largely unattainable if their central mechanisms of action remain unknown. The objective of this study is to elucidate the primary determinants of clinical response to a novel oral medication, sodium oxybate (Xyrem®), in alcohol-responsive SD and VT patients. Using a comprehensive approach of clinico-behavioral testing, neuroimaging and pharmacogenetics, we aim to determine the clinical response of SD and VT symptoms to sodium oxybate and identify the primary markers of its clinical benefits. This study will use a controlled experimental design that focuses on detailed characterization of primary effects of a novel oral medication, sodium oxybate, for treatment of SD and VT symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with SD and combined SD and VT will have a clinically documented adductor or abductor form of disorder, either with or without positive effects of alcohol on their voice symptoms;
2. Healthy controls will be healthy volunteers with a negative history of laryngeal, neurological, or psychiatric problems (existing neuroimaging data will be used);
3. Age from 21 to 80 years.
4. Native English speakers.
5. Right-handedness (based on Edinburgh Handedness Inventory).

Exclusion Criteria:

1. Subjects who are incapable of giving an informed consent will be excluded from the study.
2. Pregnant and breastfeeding women until a time when they are no longer pregnant or breastfeeding will be excluded from the study. All patients of childbearing potential will be required to agree to use a reliable method of contraception prior to and during the study. The method of contraception will be documented in the patient's research chart. All women of childbearing potential will undergo a urine pregnancy test, which must be negative for study participation.
3. All patients with a past or present history of the following conditions will be excluded from the study;

   1. Except for SD and dystonic VT, any neurological disorders, such as stroke, movement disorders, brain tumors, traumatic brain injury with loss of consciousness, ataxias, myopathies, myasthenia gravis, demyelinating diseases, alcoholism, drug dependence. Patients with tremor affecting other body parts will be excluded from the study. All patients who have dystonic movements in the body regions other than the larynx will be excluded from the study. This will allow maintaining the homogenous patient population and evaluating central drug effects without confounding by the presence of other neurological conditions.
   2. Any psychiatric problems, such as schizophrenia, major and/or bipolar depression, obsessive-compulsive disorder, will be excluded to maintain the homogenous patient population and allow for the evaluation of central drug effect without confounding by the presence of psychiatric conditions.
   3. Any laryngeal problems, such as vocal fold paralysis, paresis, carcinoma, chronic laryngitis, will be excluded from the study.
   4. Patients with a known past or present history of grade 2 or higher hepatic and renal dysfunction according to the NCI criteria will be excluded.
   5. Patients with a known past or present history of moderate to severe congestive heart failure will be excluded.
   6. Patients with a known past or present history of cognitive impairment and active suicidal ideations will be excluded.
4. Patients who are not symptomatic due to treatment with botulinum toxin injections into the laryngeal muscles will be excluded from the study until the time when they are fully symptomatic. The duration of positive effects of botulinum toxin vary from patient to patient, lasting on average 3-4 months. All patients will be evaluated to ensure that they are fully symptomatic prior to the entering the study.
5. To avoid the possibility of confounding effects of drugs acting upon the central nervous system, all patients will be questioned about any prescribed or over-the-counter medications as part of their initial intake screening. Those patients who receive medication(s) affecting the central nervous system (except for sodium oxybate) will be excluded from the study.
6. Patients will be asked whether they have undergone any head and neck surgeries, particularly any brain surgery and laryngeal surgeries, such as thyroplasty, laryngeal denervation, and selective laryngeal adductor denervation-reinnervation. Because both brain and laryngeal surgery may potentially lead to the brain structure and function re-organization, all subjects with a history of brain and/or laryngeal surgery will be excluded from the study.
7. Patients who have tattoos, ferromagnetic objects in their bodies (e.g., implanted stimulators, surgical clips, prosthesis, artificial heart valve, etc.) that are not MRI comparable and/or cannot be removed for the purpose of MRI study participation will be excluded from the study.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2018-01-22 (Actual); Primary Completion 2021-12-29 (Actual); Study Completion 2024-10-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristina Simonyan, MD, PhD, Principal Investigator — Massachusetts Eye and Ear
Locations (1):
- Massachusetts Eye and Ear, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Simonyan K, Frucht SJ. Long-term Effect of Sodium Oxybate (Xyrem(R)) in Spasmodic Dysphonia with Vocal Tremor. Tremor Other Hyperkinet Mov (N Y). 2013 Dec 9;3:tre-03-206-4731-1. doi: 10.7916/D8CJ8C5S. eCollection 2013. PMID 24386608
- [Background] Rumbach AF, Blitzer A, Frucht SJ, Simonyan K. An open-label study of sodium oxybate in Spasmodic dysphonia. Laryngoscope. 2017 Jun;127(6):1402-1407. doi: 10.1002/lary.26381. Epub 2016 Nov 3. PMID 27808415
- [Background] Battistella G, Fuertinger S, Fleysher L, Ozelius LJ, Simonyan K. Cortical sensorimotor alterations classify clinical phenotype and putative genotype of spasmodic dysphonia. Eur J Neurol. 2016 Oct;23(10):1517-27. doi: 10.1111/ene.13067. Epub 2016 Jun 27. PMID 27346568
- [Background] Kirke DN, Battistella G, Kumar V, Rubien-Thomas E, Choy M, Rumbach A, Simonyan K. Neural correlates of dystonic tremor: a multimodal study of voice tremor in spasmodic dysphonia. Brain Imaging Behav. 2017 Feb;11(1):166-175. doi: 10.1007/s11682-016-9513-x. PMID 26843004
- [Background] Kirke DN, Frucht SJ, Simonyan K. Alcohol responsiveness in laryngeal dystonia: a survey study. J Neurol. 2015 Jun;262(6):1548-56. doi: 10.1007/s00415-015-7751-2. Epub 2015 May 1. PMID 25929664
- [Background] Simonyan K, Ludlow CL. Abnormal activation of the primary somatosensory cortex in spasmodic dysphonia: an fMRI study. Cereb Cortex. 2010 Nov;20(11):2749-59. doi: 10.1093/cercor/bhq023. Epub 2010 Mar 1. PMID 20194686
- See also: NIH grant description — https://reporter.nih.gov/search/dPfQ17fnGUOqdn2Teo9Xwg/project-details/10240318

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted between January 22, 2018, and December 29, 2021. The COVID-19 pandemic and the associated lockdown of human research activities fully paused patient recruitment and the conduct of study procedures between March 2020 and December 2020.
Pre-assignment Details: Pre-specified to LD patients with and without dystonic voice tremor regardless of alcohol responsiveness of symptoms.
  9 patients were excluded because of a history of suicidal ideations (n= 3), absence of symptoms at the time of study participation (n= 3), left-handedness (n= 1), presence of multifocal dystonia (n= 1), and contraindications to MRI (n= 1).
Groups:
- Laryngeal Dystonia With and Without Dystonic Tremor of Voice: Sodium Oxybate, Then Placebo: Participants with alcohol-responsive and non-responsive LD with/without dystonic tremor of voice first received a single dose of oral solution of sodium oxybate 1.5 g. After a 24-hour washout period, they then received oral solution of placebo (matching sodium oxybate 1.5 g).
  According to a priori hypothesis, the analysis was conducted based on the alcohol-responsiveness of symptoms, regardless of period sequence.
  Baseline measures are described based on LD phenotype and alcohol-responsiveness for detailed cohort description.
- Laryngeal Dystonia With and Without Dystonic Tremor of Voice: Placebo, Then Sodium Oxybate: Participants with alcohol-responsive and non-responsive LD with/without dystonic tremor of voice first received a single dose of oral solution of placebo (matching sodium oxybate 1.5 g). After a 24-hour washout period, they then received oral solution of sodium oxybate 1.5 g.
  According to a priori hypothesis, the analysis was conducted based on the alcohol-responsiveness of symptoms, regardless of period sequence.
  Baseline measures are described based on LD phenotype and alcohol-responsiveness for detailed cohort description.
Period: Period 1
Arm/Group | Laryngeal Dystonia With and Without Dystonic Tremor of Voice: Sodium Oxybate, Then Placebo | Laryngeal Dystonia With and Without Dystonic Tremor of Voice: Placebo, Then Sodium Oxybate
Started | 55 | 53
Completed | 53 | 53
Not Completed | 2 | 0
Not completed — Adverse Event | 2 | 0
Period: Period 2
Arm/Group | Laryngeal Dystonia With and Without Dystonic Tremor of Voice: Sodium Oxybate, Then Placebo | Laryngeal Dystonia With and Without Dystonic Tremor of Voice: Placebo, Then Sodium Oxybate
Started | 53 | 53
Completed | 53 | 53
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Pre-specified to analysis based only on the diagnosis (LD, LD/DTv) and alcohol responsiveness (EtOH+, EtOH-).
Groups:
- (1) Alcohol-responsive (EtOH+) Laryngeal Dystonia; (2) Alcohol-responsive (EtOH+) Laryngeal Dystonia With Dystonic Tremor of Voice: For analysis, patients in groups (1) Alcohol-responsive (EtOH+) Laryngeal Dystonia and (2) Alcohol-responsive (EtOH+) Laryngeal Dystonia with Dystonic Tremor of Voice were combined into the overall EtOH+ group.
- (3) Alcohol-non-responsive (EtOH-) Laryngeal Dystonia; (4) Alcohol-non-responsive (EtOH-) Laryngeal Dystonia With Dystonic Tremor of Voice: For analysis, patients in groups (3) Alcohol-non-responsive (EtOH-) Laryngeal Dystonia and (4) Alcohol-non-responsive (EtOH-) Laryngeal Dystonia with Dystonic Tremor of Voice were combined into the overall EtOH- group.
- Total: Total of all reporting groups
Arm/Group | (1) Alcohol-responsive (EtOH+) Laryngeal Dystonia | (2) Alcohol-responsive (EtOH+) Laryngeal Dystonia With Dystonic Tremor of Voice | (3) Alcohol-non-responsive (EtOH-) Laryngeal Dystonia | (4) Alcohol-non-responsive (EtOH-) Laryngeal Dystonia With Dystonic Tremor of Voice | Total
Number analyzed (Participants) | 23 | 29 | 30 | 26 | 108
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 19 | 16 | 23 | 12 | 70
  >=65 years | 4 | 13 | 7 | 14 | 38
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 56.0 [48.5 to 61.5] | 62.0 [52.0 to 68.0] | 57.0 [48.0 to 63.8] | 66.5 [54.3 to 71.8] | 59.5 [50.0 to 68.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 26 | 17 | 18 | 76
  Male | 8 | 3 | 13 | 8 | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 23 | 29 | 30 | 26 | 108
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 1 | 1 | 2 | 7
  White | 20 | 28 | 29 | 24 | 101
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Handedness [Count of Participants; unit: Participants]
  Right-handed | 23 | 29 | 30 | 26 | 108
  Left-handed | 0 | 0 | 0 | 0 | 0
Monolingual native English Language [Count of Participants; unit: Participants] | 23 | 29 | 30 | 26 | 108
Cognitive function [Count of Participants; unit: Participants] — Montreal Cognitive Assessment Test Score
  Participants
    ≥ 26 points (normal cognitive function) | 23 | 29 | 30 | 26 | 108
    < 26 points (impaired cognitive function) | 0 | 0 | 0 | 0 | 0
Dystonia phenotype [Count of Participants; unit: Participants]
  Adductor type | 12 | 13 | 17 | 16 | 58
  Abductor type | 10 | 12 | 12 | 9 | 43
  Mixed adductor and abductor type | 1 | 4 | 1 | 1 | 7
Family history of dystonia [Count of Participants; unit: Participants]
  Familial type | 3 | 2 | 2 | 1 | 8
  Sporadic type | 20 | 27 | 28 | 25 | 100
Age of onset [Median (Inter-Quartile Range); unit: years] | 38.0 [31.5 to 46.0] | 50.0 [32.0 to 56.0] | 43.5 [32.5 to 52.8] | 46.5 [31.0 to 60.0] | 44.0 [31.8 to 54.0]
Dystonia duration [Median (Inter-Quartile Range); unit: years] | 13.0 [9.5 to 20.0] | 13.0 [8.0 to 22.0] | 11.0 [5.3 to 23.5] | 13.4 [7.3 to 28.0] | 13.0 [7.0 to 22.0]
Botulinum toxin treatment [Count of Participants; unit: Participants] | 20 | 26 | 26 | 21 | 93
Centrally acting medications [Count of Participants; unit: Participants] | 4 | 8 | 7 | 5 | 24

OUTCOME MEASURES:

1. Primary Outcome: Symptom Severity
Description: A combined clinician-objective and patient-subjective change in visual analog scale (min-max 0-100, a higher score is the worse outcome) score of symptom severity before and after drug vs. placebo intake.
  For analysis, patients in groups (1) Alcohol-responsive (EtOH+) Laryngeal Dystonia and (2) Alcohol-responsive (EtOH+) Laryngeal Dystonia with Dystonic Tremor of Voice were combined into the overall EtOH+ group.
  For analysis, patients in groups (3) Alcohol-non-responsive (EtOH-) Laryngeal Dystonia and (4) Alcohol-non-responsive (EtOH-) Laryngeal Dystonia with Dystonic Tremor of Voice were combined into the overall EtOH- group.
Time Frame: 40 min after drug or placebo administration
Measure: Least Squares Mean (98.75% Confidence Interval); unit: score on a scale
Groups:
- Alcohol-responsive (EtOH+) Laryngeal Dystonia; Alcohol-non-responsive (EtOH-) Laryngeal Dystonia: Laryngeal dystonia with and without dystonic tremor of voice
Arm/Group | Alcohol-responsive (EtOH+) Laryngeal Dystonia | Alcohol-non-responsive (EtOH-) Laryngeal Dystonia
Number analyzed (Participants) | 50 | 56
score on a scale
  Sodium oxybate | 28.0 [21.0 to 35.0] | 18.6 [12.0 to 25.2]
  Placebo | 14.2 [7.2 to 21.2] | 12.3 [5.7 to 19.0]
Statistical Analysis 1: Comparison: Alcohol-responsive (EtOH+) Laryngeal Dystonia vs Alcohol-non-responsive (EtOH-) Laryngeal Dystonia; Test type: Superiority — The primary efficacy outcome was analyzed using a restricted maximum likelihood (REML)-based linear mixed-effect model. The analysis included group, treatment, and treatment period as interacting fixed effects and subject as random effect. An unstructured covariance structure was used to model the within-patient errors; p = 0.01, Mixed Models Analysis

2. Primary Outcome: Minimum Treatment Efficacy
Description: Pre-specified to analysis based only on alcohol responsiveness (EtOH+). A combined clinician-objective and patient-subjective change in visual analog scale score (min-max 0-100, a higher score is the worse outcome) of symptom severity in EtOH+ patients.
Time Frame: 40 min after drug or placebo administration
Population: Pre-specified to only report Alcohol-responsive (EtOH+) Laryngeal Dystonia Arm
Measure: Mean (98.75% Confidence Interval); unit: percentage of symptom change
Groups:
- Alcohol-responsive (EtOH+) Laryngeal Dystonia: Laryngeal dystonia with and without dystonic tremor of voice. Pre-specified to analysis based only on alcohol responsiveness (EtOH+).
Arm/Group | Alcohol-responsive (EtOH+) Laryngeal Dystonia
Number analyzed (Participants) | 50
percentage of symptom change
  Symptom improvement ≥ 16%: number analyzed (Participants) | 32
  Symptom improvement ≥ 16% | 40.81 [34.7 to 48.6]
  Symptom improvement < 16%: number analyzed (Participants) | 18
  Symptom improvement < 16% | 4.76 [1.1 to 8.1]
Statistical Analysis 1: Comparison: Alcohol-responsive (EtOH+) Laryngeal Dystonia; The minimum and average efficacy of sodium oxybate vs. placebo in improving symptoms compared to the baseline were determined using binomial logistic regression; Test type: Other — The minimum and average efficacy (in % symptom change) of sodium oxybate versus placebo in improving symptoms compared to the baseline was determined using binomial logistic regression; p = 0.05, Regression, Logistic

3. Secondary Outcome: Treatment Efficacy Dependent on LD Clinical Type
Description: A combined clinician-objective and patient-subjective change in visual analog scale (min-max 0-100, a higher score is the worse outcome) score of symptom severity before and after drug vs. placebo intake.
  EtOH+ and EtOH- were stratified based on phenotypical characteristics, including LD, LD with Dystonic Tremor of Voice, Abductor LD, Adductor LD.
Time Frame: 40 min after drug or placebo administration
Measure: Mean (Standard Error); unit: score on a scale
Groups:
- Alcohol-responsive (EtOH+) Laryngeal Dystonia; Alcohol-non-responsive (EtOH-) Laryngeal Dystonia: Laryngeal dystonia
- Alcohol-responsive (EtOH+) Laryngeal Dystonia With Dystonic Tremor of Voice; Alcohol-non-responsive (EtOH-) Laryngeal Dystonia With Dystonic Tremor of Voice: Laryngeal dystonia with dystonic tremor of voice
- Alcohol-responsive Adductor Type of Laryngeal Dystonia; Alcohol-non-responsive Adductor Type of Laryngeal Dystonia: Laryngeal dystonia, adductor type
- Alcohol-responsive Abductor Type of Laryngeal Dystonia; Alcohol-non-responsive Abductor Type of Laryngeal Dystonia: Laryngeal dystonia, abductor type
Arm/Group | Alcohol-responsive (EtOH+) Laryngeal Dystonia | Alcohol-responsive (EtOH+) Laryngeal Dystonia With Dystonic Tremor of Voice | Alcohol-non-responsive (EtOH-) Laryngeal Dystonia | Alcohol-non-responsive (EtOH-) Laryngeal Dystonia With Dystonic Tremor of Voice | Alcohol-responsive Adductor Type of Laryngeal Dystonia | Alcohol-responsive Abductor Type of Laryngeal Dystonia | Alcohol-non-responsive Adductor Type of Laryngeal Dystonia | Alcohol-non-responsive Abductor Type of Laryngeal Dystonia
Number analyzed (Participants) | 23 | 27 | 30 | 26 | 25 | 20 | 33 | 21
score on a scale
  Sodium oxybate | 24.65 (4.45) | 30.54 (4.29) | 18.30 (3.07) | 18.96 (3.49) | 31.70 (5.08) | 24.85 (3.92) | 21.36 (2.86) | 14.96 (4.04)
  Placebo | 18.07 (3.99) | 10.85 (5.90) | 10.34 (1.94) | 14.47 (1.93) | 13.59 (6.07) | 13.10 (4.62) | 13.07 (1.54) | 11.32 (2.83)
Statistical Analysis 1: Comparison: Alcohol-responsive (EtOH+) Laryngeal Dystonia vs Alcohol-responsive (EtOH+) Laryngeal Dystonia With Dystonic Tremor of Voice vs Alcohol-non-responsive (EtOH-) Laryngeal Dystonia vs Alcohol-non-responsive (EtOH-) Laryngeal Dystonia With Dystonic Tremor of Voice vs Alcohol-responsive Adductor Type of Laryngeal Dystonia vs Alcohol-responsive Abductor Type of Laryngeal Dystonia vs Alcohol-non-responsive Adductor Type of Laryngeal Dystonia vs Alcohol-non-responsive Abductor Type of Laryngeal Dystonia; Test type: Other; p = 0.01, t-test, 2 sided; Mean Difference (Final Values) = 98.75

4. Secondary Outcome: Length of Treatment Efficacy
Description: The length of treatment efficacy in each EtOH+ and EtOH- group was assessed at 40, 180, and 300 min after drug vs. placebo intake compared to the baseline using a combined clinician-objective and patient-subjective change in visual analog scale (min-max 0-100, a higher score is the worse outcome) score of symptom severity.
  For analysis, patients in groups (1) Alcohol-responsive (EtOH+) Laryngeal Dystonia and (2) Alcohol-responsive (EtOH+) Laryngeal Dystonia with Dystonic Tremor of Voice were combined into the overall EtOH+ group.
  For analysis, patients in groups (3) Alcohol-non-responsive (EtOH-) Laryngeal Dystonia and (4) Alcohol-non-responsive (EtOH-) Laryngeal Dystonia with Dystonic Tremor of Voice were combined into the overall EtOH- group.
Time Frame: 40 min to 5 hours after drug or placebo administration
Population: Pre-specified to only report based on alcohol-responsiveness (EtOH+, EtOH-)
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Alcohol-responsive (EtOH+) Laryngeal Dystonia | Alcohol-non-responsive (EtOH-) Laryngeal Dystonia
Number analyzed (Participants) | 50 | 56
score on a scale
  Sodium oxybate: 40 min | 28.0 (3.06) | 18.60 (2.31)
  Sodium oxybate: 180 min | 18.63 (3.36) | 12.67 (2.40)
  Sodium oxybate: 300 min | 15.47 (4.32) | 8.33 (1.98)
  Placebo: 40 min | 14.23 (3.71) | 12.34 (1.39)
  Placebo: 180 min | 9.26 (3.61) | 9.31 (1.99)
  Placebo: 300 min | 10.30 (3.15) | 8.16 (1.84)
Statistical Analysis 1: Comparison: Alcohol-responsive (EtOH+) Laryngeal Dystonia vs Alcohol-non-responsive (EtOH-) Laryngeal Dystonia; Test type: Other; p = 0.01, ANOVA

5. Secondary Outcome: Relationship Between Alcohol-responsiveness of Symptoms and Drug-induced Symptom Improvement
Description: A combined clinician-objective and patient-subjective change in visual analog scale (min-max 0-100, a higher score is the worse outcome) score of symptom severity before and 40 min after drug vs. placebo intake.
  For analysis, patients in groups (1) Alcohol-responsive (EtOH+) Laryngeal Dystonia and (2) Alcohol-responsive (EtOH+) Laryngeal Dystonia with Dystonic Tremor of Voice were combined into the overall EtOH+ group.
  For analysis, patients in groups (3) Alcohol-non-responsive (EtOH-) Laryngeal Dystonia and (4) Alcohol-non-responsive (EtOH-) Laryngeal Dystonia with Dystonic Tremor of Voice were combined into the overall EtOH- group.
Time Frame: 40 min after drug or placebo administration
Population: Pre-specified to only report based on alcohol-responsiveness (EtOH+, EtOH-)
Measure: Number (98.75% Confidence Interval); unit: correlation coefficient
Arm/Group | Alcohol-responsive (EtOH+) Laryngeal Dystonia | Alcohol-non-responsive (EtOH-) Laryngeal Dystonia
Number analyzed (Participants) | 50 | 56
correlation coefficient
  Sodium oxybate | 0.45 [0.10 to 6.88] | 0.09 [-0.024 to 0.35]
  Placebo | 0.06 [-0.034 to 0.39] | 0.22 [-0.10 to 0.55]
Statistical Analysis 1: Comparison: Alcohol-responsive (EtOH+) Laryngeal Dystonia vs Alcohol-non-responsive (EtOH-) Laryngeal Dystonia; Test type: Other; p = 0.01, Pearson correlation

6. Secondary Outcome: Relationship Between Symptom Severity Change and Dystonia Clinical Characteristics
Description: as for outcome 5
Time Frame: 40 min after drug or placebo administration
Population: Pre-specified to only report based on alcohol-responsiveness (EtOH+, EtOH-)
Measure: Number (98.75% Confidence Interval); unit: correlation coefficient
Arm/Group | Alcohol-responsive (EtOH+) Laryngeal Dystonia | Alcohol-non-responsive (EtOH-) Laryngeal Dystonia
Number analyzed (Participants) | 50 | 56
correlation coefficient
  Sodium oxybate: duration | -0.17 [-0.51 to 0.16] | 0.10 [-0.26 to 0.49]
  Placebo: duration | 0.18 [-0.21 to 0.52] | 0.16 [-0.17 to 0.44]
  Sodium oxybate: age of symptom onset | 0.16 [-0.14 to 0.47] | -0.15 [-0.43 to 0.18]
  Placebo: age of symptom onset | -0.18 [-0.46 to 0.22] | -0.09 [-0.40 to 0.30]
  Sodium oxybate: baseline symptom severity | -0.05 [-0.31 to 0.20] | -0.04 [-0.47 to 0.36]
  Placebo: baseline symptom severity | 0.24 [-0.20 to 0.58] | -0.11 [-0.39 to 0.18]
Statistical Analysis 1: Comparison: Alcohol-responsive (EtOH+) Laryngeal Dystonia vs Alcohol-non-responsive (EtOH-) Laryngeal Dystonia; Test type: Other; p = 0.01, Pearson correlation

ADVERSE EVENTS:
Time Frame: 5 hours and a 24-hour follow-up
Description: Safety was documented as a change from baseline in vital signs (blood pressure, pulse rate), cognitive function (MoCA), suicidality (C-SSRS), and daytime sleepiness (Epworth sleepiness scale). Adverse events were assessed using a structured side effects questionnaire and unstructured patient reporting (unprompted self-reporting by patients) as none, mild, moderate, or severe.
  Pre-specified to report adverse events by alcohol responsiveness and intervention only.
Groups:
- Sodium Oxybate: Alcohol-responsive (EtOH+) Laryngeal Dystonia; Placebo: Alcohol-responsive (EtOH+) Laryngeal Dystonia: For analysis, patients in groups (1) Alcohol-responsive (EtOH+) Laryngeal Dystonia and (2) Alcohol-responsive (EtOH+) Laryngeal Dystonia with Dystonic Tremor of Voice were combined into the overall EtOH+ group.
- Sodium Oxybate: Alcohol-non-responsive (EtOH-) Laryngeal Dystonia; Placebo: Alcohol-non-responsive (EtOH-) Laryngeal Dystonia: For analysis, patients in groups (3) Alcohol-non-responsive (EtOH-) Laryngeal Dystonia and (4) Alcohol-non-responsive (EtOH-) Laryngeal Dystonia with Dystonic Tremor of Voice were combined into the overall EtOH- group.
Arm/Group | Sodium Oxybate: Alcohol-responsive (EtOH+) Laryngeal Dystonia | Placebo: Alcohol-responsive (EtOH+) Laryngeal Dystonia | Sodium Oxybate: Alcohol-non-responsive (EtOH-) Laryngeal Dystonia | Placebo: Alcohol-non-responsive (EtOH-) Laryngeal Dystonia
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/50 | 0/56 | 0/56
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50 | 0/56 | 0/56
Other Adverse Events (participants affected / at risk) | 29/50 | 8/50 | 37/56 | 13/56
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sodium Oxybate: Alcohol-responsive (EtOH+) Laryngeal Dystonia (N=50) | Placebo: Alcohol-responsive (EtOH+) Laryngeal Dystonia (N=50) | Sodium Oxybate: Alcohol-non-responsive (EtOH-) Laryngeal Dystonia (N=56) | Placebo: Alcohol-non-responsive (EtOH-) Laryngeal Dystonia (N=56)
Mild Dizziness/ lightheadedness/unsteadiness/clumsiness (Nervous system disorders) | 24 | 4 | 27 | 8
Mild Blurred vision (Nervous system disorders) | 2 | 1 | 4 | 0
Mild Headache (Nervous system disorders) | 4 | 2 | 3 | 2
Mild Trouble concentrating (Nervous system disorders) | 3 | 0 | 1 | 1
Mild Confusion (Nervous system disorders) | 1 | 0 | 0 | 0
Mild Restlessness (Nervous system disorders) | 0 | 0 | 1 | 0
Mild Disorientation (Nervous system disorders) | 0 | 0 | 1 | 1
Mild Depression (Nervous system disorders) | 1 | 0 | 0 | 0
Mild Feeling hangover (Nervous system disorders) | 0 | 0 | 1 | 0
Mild Nervousness (Nervous system disorders) | 0 | 1 | 0 | 0
Mild Lethargy (Nervous system disorders) | 0 | 0 | 0 | 1
Mild Nausea (Gastrointestinal disorders) | 1 | 0 | 8 | 1
Mild Dry mouth (Gastrointestinal disorders) | 3 | 3 | 3 | 1
Mild Vomiting (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Mild Diarrhea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Mild Stomach pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Mild Daytime sleepiness (Nervous system disorders) | 10 | 3 | 8 | 0
Moderate Dizziness/ lightheadedness/unsteadiness/clumsiness (Nervous system disorders) | 1 | 0 | 2 | 0
Moderate Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
A single-center trial: However, the patients were recruited across the US, the UK, and Australia, thus expanding the generalizability of the findings.

An inclusion of a greater number of Non-Hispanic White females: LD is well-documented to affect the Non-Hispanic White population with a 4:1 female to male prevalence. Thus, the demographics of patients recruited for this trial reflect the clinical demographics of the disorder in general.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2024-03-04): https://cdn.clinicaltrials.gov/large-docs/58/NCT03292458/Prot_SAP_ICF_002.pdf